CLINICAL TRIAL: NCT00379600
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Investigate the Anti-inflammatory and Metabolic Effects of Rosiglitazone XR, 8mg Once Daily, in Subjects With Rheumatoid Arthritis
Brief Title: The Anti-Inflammatory And Metabolic Effects Of Rosiglitazone In Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARA102198
Record Dates: First submitted 2006-09-21; First posted 2006-09-22 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Arthritis, Rheumatoid
Keywords: Anti-inflammatory treatment; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: rosiglitazone XR

SUMMARY:
To assess whether the anti-inflammatory effects of rosiglitazone result in improvements in Rheumatoid Arthritis symptoms in patients for whom their existing Disease Modifying Anti-Rheumatic Drug (DMARD) treatment does not give adequate relief.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid Arthritis insufficiently controlled by existing disease-modifying anti-rheumatic drugs
* Subjects will have at least 6 swollen joints plus 2 of the following: 6 tender joints (of 28 joints); early morning stiffness lasting more than 30 minutes; ESR greater or equal to 28mm/h
* must be receiving a stable dose of disease-modifying anti-rheumatic therapy for at least 2 months prior to participating in the study.

Exclusion criteria:

* Women who are lactating, pregnant, or planning to become pregnant during the course of the study including 30 days following conclusion of study medication
* Systolic blood pressure (SBP) >165 mmHg or diastolic blood pressure (DBP) >95 mmHg while receiving optimal antihypertensive therapy
* Any clinically significant abnormality identified on the screening physical exam, laboratory tests, or ECG, which in the judgement of the Investigator makes the subject unsuitable for inclusion in the study
* a history of alcohol abuse within the past 3 years or consumes >3 units per day for males and >2 units per day for females or has a history of cirrhosis or stigmata of chronic liver disease
* a history of liver disease or has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels >2.5 times upper limit of normal and total bilirubin levels greater than 1.5 times the upper limit of normal (unless associated with predominantly indirect bilirubin or Gilbert's syndrome) at screening
* using glucocorticoid at doses >10 mg/day currently or within the last 3 months or may be expected to do so during the course of the study
* The subject's dose of NSAIDs, COX-2 inhibitors or glucocorticoids has changed at any time during the past 2 weeks prior to screening or may be expected to change during the course of the study
* The subject's dose or treatment with a statin has changed at any time during the past 3 months prior to screening or may be expected to change during the course of the study
* a history of renal disease or has serum creatinine = 132mol/L for males and =130mol for females
* has diabetes mellitus that requires medication or hyperglycaemia with a HbA1c of >7%
* History of new cardiovascular event within the last 6 months (i.e., intervention, percutaneous coronary intervention, vascular surgery, acute coronary syndrome [non Q-wave myocardial infarction, Q-wave myocardial infarction, unstable angina) or significant arrhythmia; or major intervention (e.g., cardiac surgery or angiography plus stenting) scheduled
* Concurrent or past medical history of congestive heart failure or pulmonary oedema
* A presence of severe peripheral oedema or a medically serious fluid-related event
* has significant cardiac, pulmonary, metabolic, renal, hepatic, gastrointestinal or immunological conditions that, in the opinion of the Investigator and/or GSK medical monitor, places the subject at an unacceptable risk as a participant in this trial
* a history of malignancy in the last 5 years, except for surgically cured basal cell carcinoma (>2 years prior to first dosing)
* a history of HIV, or chronic hepatitis B or positive C serology
* a history of drug abuse
* has participated in a clinical trial within the 3 months before the start of the study for non-biological therapy; or within 6 months of a biological therapy
* on a biological therapy or has received biological therapy within 6 months prior to screening
* has donated blood in excess of 500 mL within 56 days prior to dosing
* The subject is at risk of non-compliance in following directions or adhering to study restrictions
* a history of drug or other allergy, which, in the opinion of the physician responsible, contraindicates their participation
* has anaemia defined by haemoglobin concentration <11 g/dL for males or <10 g/dL for females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2004-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Disease Activity Score (DAS) following 6 months of treatment | 6 Months

SECONDARY OUTCOMES:
Disease activity at 3 months and 6 months, e.g., number of affected joints Patient Assessments of Improvements in Disease Activity, e.g., fatigue and pain assessment Assessment of safety, tolerability and biological activity | Disease activity at 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Lithuania (2):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Vilnius
- GSK Investigational Site, Glasgow, Lanarkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: ARA102198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: ARA102198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: ARA102198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: ARA102198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: ARA102198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: ARA102198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: ARA102198 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register